CLINICAL TRIAL: NCT05845281
Title: Comparison of Erector Spina Plane Block and Intravenous Patient-controlled Analgesia in Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Comparison of Erector Spinae Plane Block and Intravenous Patient-controlled Analgesia in Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Hacı Yusuf Güneş, MD, Assistant proffesor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02.03. 2022/04
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Nephrolithiasis; Percutaneous; Analgesia; PCA
Keywords: Percutaneous; Nephrolithotomy; Plane Block; Patient-controlled analgesia
MeSH Terms: conditions — Nephrolithiasis; Agnosia | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: The patients weredivided in two groups. Thirty patients were assigned to each group. Standard general anesthesia procedure was applied to all patients. Perioperative hemodynamic monitoring was performed. Group ESP underwent an erector spina block after the surgical procedure. Intravenous patient-controlled analgesia with tramadol was applied to group PCA patients. VAS score, need for additional analgesia, patient satisfaction (Likert scale), mobilization times and vital signs were recorded at 30 minutes, 1th, 3th, 6th and 12th hours after the operation.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESP, Erector Spina Plane Block (n= 30) (Active Comparator): After the surgical procedure was completed in patients who underwent general anesthesia, the necessary sterility was provided for the ESPB procedure while the patient was in the lateral position. 1mg/kg 0.5% bupivacaine + 1mg/kg 2% lidocaine was drawn into the same syringe and the volume was completed to 20 ml with normal saline. A linear 10-18 MHz USG probe was placed at the thoracic 7 level (Esaote MyLab 30, Geneva, Italy) in the paramedian plane between two transverse processes. The prepared local anesthetic drug was administered under the guidance of USG.
  Interventions: Procedure: Bupivakain + deksametazon Adjuvant
- Group PCA, Patient Controlled Analgesia (n= 30) (Experimental): For patients in the PCA group, 200 mg of tramadol was placed in 100cc of 0.9% NaCl. Set to PCA device. A 50mg loading dose was administered 10 minutes before the patient was extubated. After extubating, a bolus dose of 20 mg was started, with a 30-minute lock-in time, and an infusion dose of 5mg/hour. The 4-hour maximum limit was set to 200 mg.
  Interventions: Procedure: Bupivakain + deksametazon Adjuvant

INTERVENTIONS:
Procedure: Bupivakain + deksametazon Adjuvant — In patients who underwent general anesthesia, after the surgical procedure was completed, after sterility was ensured for the ESP group while the patient was in the lateral position for the ESPB procedure, the linear 10-18 MHz USG probe (Esaote MyLab 30, Geneva, Italy) was placed between two transverse processes in the paramedian plane and increased from 1mg/kg to %1 at the T7 level. 20 ml of 0.5 bupivacaine (Buvasin®, Vem, Istanbul, Turkey) + 2% arrhythmic residual SF from 1mg/kg was administered. For patients in the PCA group, 200 mg of tramadol was placed in 100cc of 0.9% NaCl. Set to PCA device. A 50mg loading dose was administered 10 minutes before the patient was extubated. After extubating, a bolus dose of 20 mg was started, with a 30-minute lock-in time, and an infusion dose of 5mg/hour. The 4-hour maximum limit was set to 200 mg.
  Other Names: PCA, Patient Controlled Analgesia

SUMMARY:
The primary purpose of this study was to compare the effects of erector spinal plane block (ESP) and IV patient-controlled analgesia (PCA) performed to provide analgesia in percutaneous nephrolithotomy surgeries on visual analog skala (VAS), additional analgesia need, patient satisfaction and mobilization times.

DETAILED DESCRIPTION:
ASA I-III patients aged 18-65 years who underwent percutaneous nephrolithotomy at Van Yüzüncü Yıl University Faculty of Medicine were included in the study.

The patients were informed about the study during the preoperative evaluation. In the randomized single-blind closed-envelope study, 30 patients ineach group and a total of 60 patients were included. Standard general anesthesia procedure was applied to all patients. Standard general anesthesia procedure was applied to all patients. Perioperative hemodynamic monitoring was performed. In patients who underwent general anesthesia, after the surgical procedure was completed, after sterility was ensured for the ESP group while the patient was in the lateral position for the ESPB procedure, the linear 10-18 MHz USG probe (Esaote MyLab 30, Geneva, Italy) was placed between two transverse processes in the paramedian plane and increased from 1mg/kg to %1 at the T7 level. 20 ml of 0.5 bupivacaine (Buvasin®, Vem, Istanbul, Turkey) + 2% arrhythmic residual SF from 1mg/kg was administered. For patients in the PCA group, 200 mg of tramadol was placed in 100cc of 0.9% NaCl. Set to PCA device. A 50mg loading dose was administered 10 minutes before the patient was extubated. After extubating, a bolus dose of 20 mg was started, with a 30-minute lock-in time, and an infusion dose of 5mg/hour. The 4-hour maximum limit was set to 200 mg.

VAS score, need for additional analgesia, patient satisfaction (Likert scale), mobilization times and vital signs were recorded at 30 minutes, p1, 3, 6 and 12 hours after the operation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) class I-III,
* Between 18-65 years old,
* Percutaneous nephrolithotomy surgery,
* Patients who agreed to participate in the study

Exclusion Criteria:

* Obesity (BMI≥ 35)
* Coagulopathy
* Active Infection
* Drug allergies
* Pregnancy
* 65 years and older

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
Post operative analgesia | 24 hours
  Visual Analog Scale score were recorded at the post operative 30 minutes, 1st, 3rd, 6th and 12th hours after the operation. High VAS score was interpreted as severe pain in patients. When the VAS score was 4 and above, additional analgesic (15 mg/kg paracetamol) was given intravenously.
Additional analgesic drug | 24 hours
  When the VAS score was 4 and above, 15 mg/kg paracetamol was given intravenously. Additional analgesic drug (Paracetamol) was recorded in milligrams.
Patient satisfaction | 24 hours
  Patient satisfaction was recorded using a Likert scale at the 30th minute, 1st, 3rd, 6th and 12th hours after the operation.
  Patient satisfaction was scored between 1 and 5 using a Likert scale at the 30th minute, 1st, 3rd, 6th and 12th hours postoperatively. 1 point not satisfied at all, 2 points dissatisfied, 3 points not sure, 4 points satisfied, 5 points very satisfied.
First walking time after surgery | 24 hours
  Mobilization status was checked and recorded at the 30th minute, 1st, 3rd, 6th and 12th hours after the surgery. We accepted the extubation time as the postoperative 0th hour. We determined the time when the patients started walking for the first time after the surgery accordingly.

CONTACTS AND LOCATIONS:
Overall Officials: Hacı Yusuf YG Güneş, Assist.prof, Principal Investigator — Van Yüzüncü Yıl University Van, Turkey
Locations (1):
- Haci Yusuf GUNES, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be share for other resarchers.
Supporting Information: Study Protocol, SAP
Time Frame: 6 month
Access Criteria: The access can be provided via the e-mail addresses below hyusufgunes@hotmail.com

REFERENCES:
- [Background] Liu Y, Zhu W, Zeng G. Percutaneous nephrolithotomy with suction: is this the future? Curr Opin Urol. 2021 Mar 1;31(2):95-101. doi: 10.1097/MOU.0000000000000854. PMID 33470685
- [Background] Zeng G, Cai C, Duan X, Xu X, Mao H, Li X, Nie Y, Xie J, Li J, Lu J, Zou X, Mo J, Li C, Li J, Wang W, Yu Y, Fei X, Gu X, Chen J, Kong X, Pang J, Zhu W, Zhao Z, Wu W, Sun H, Liu Y, la Rosette J. Mini Percutaneous Nephrolithotomy Is a Noninferior Modality to Standard Percutaneous Nephrolithotomy for the Management of 20-40mm Renal Calculi: A Multicenter Randomized Controlled Trial. Eur Urol. 2021 Jan;79(1):114-121. doi: 10.1016/j.eururo.2020.09.026. Epub 2020 Sep 29. PMID 32994063
- [Background] Deng W, Hou XM, Zhou XY, Zhou QH. Rhomboid intercostal block combined with sub-serratus plane block versus rhomboid intercostal block for postoperative analgesia after video-assisted thoracoscopic surgery: a prospective randomized-controlled trial. BMC Pulm Med. 2021 Feb 25;21(1):68. doi: 10.1186/s12890-021-01432-7. PMID 33632189